CLINICAL TRIAL: NCT07015203
Title: The Combined First Trimester Screening
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: University Hospital Olomouc (Other); Institute for the Care of Mother and Child, Prague, Czech Republic (Other); Krajská zdravotní, a.s. - Nemocnice Most, o.z. (Other)
Responsible Party: Sponsor
Other Study IDs: UZIS 2025/4
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Preeclampsia (PE); Fetal Growth Restriction; Congenital Abnormalities; Preterm Labor; Intrauterine Fetal Demise; Genetics Syndrome; Pregnancy Overdue - Week 41+6
Keywords: preeclampsia; prediction; prevention; maternal risk factors; Mean Arterial Pressure; Uterine artery Pulsatility Index; Placental Growth Factor; acetylsalicylic acid; Czech Republic
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Congenital Abnormalities; Obstetric Labor, Premature; Stillbirth; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A woman over 18 years old in the first trimester of pregnancy (11th-13th gestational week): A participant in the project must have signed the Consent to Participate in the Project and the Consent to the Processing of Personal Data.

SUMMARY:
The project is a national, prospective, multicenter pilot project. The project is focus on setting up the combined first trimester screening in the Czech Republic.

The combined first trimester screening is aimed at predicting and detecting the most serious obstetric complications, such as the great obstetrical syndromes (preeclampsia, fetal growth restriction, preterm labor and intrauterine fetal demise "IUFD") and structural congenital defects (morphological and chromosomal).

The primary objective of the project is to create a unified methodology for performing and evaluating the combined first trimester screening in connection with the National Health Information System (hereinafter referred to as "NHIS"), which will enable recording, providing analysis and linking recorded clinical parameters with data in the NHIS. The pilot project will also provide data for modeling appropriate mechanisms for reimbursement from public health insurance.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter pilot project. The project is focus on setting up the combined first trimester screening in the Czech Republic.

The global goal of the project is to develop and implement an appropriate care system for pregnant women, specifically by unifying (standardizing) the process of assessing the fetal anomaly scan and the risk of preeclampsia. This examination in first trimester of pregnancy is not routinely covered by public health insurance and is therefore not available to all women. By standardizing and unifying the screening process, the quality and accessibility of care will be improved for all population groups. This will lead to better health outcomes for the population, including socially excluded groups.

The methodology will be tested on a sample of 2000 women in the first trimester of pregnancy.

The combined firts trimester screening will include collecting the required parameters maternal, ultrasound, biochemical and biophysical. The Fetal Medicine Foundation (FMF) certified software will be used to determine them. FMF certified software will be used to calculate/assess the individual risk of developing pre-eclampsia, fetal growth restriction and the occurrence of fetal chromosomal aneuploidies (trisomies of chromosomes 21, 18 and 13) based on the input parameters.

The project is supported by the European Social Fund Plus (Operational Program Employment plus) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0003855.

ELIGIBILITY:
Inclusion Criteria:

* A woman over 18 years old in the first trimester of pregnancy (11th-13th gestational week)
* Signed the Consent to Participate in the Project and GDPR.

Exclusion Criteria:

* Unsigned the Consent to Participate in the Project and the Consent to the Processing of Personal Data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women matching all inclusion criteria & GDPR.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of women with identified increased risk of Preeclampsia, Fetal Growth Restriction or Fetal Chromosomal Aneuploidies (trisomies of chromosomes 21, 18 and 13) | From June 2025 to October 2026

CONTACTS AND LOCATIONS:
Overall Officials: Marek Ľubušký, prof., Study Director — THE FETAL MEDICINE CENTRE, Department of Obstetrics and Gynecology, Palacky University Olomouc, Faculty of Medicine and Dentistry, University Hospital Olomouc
Locations (3):
- Czechia (3):
  - Regional Health Corpotarion - Most Hospital, Most, Czechia
  - University Hospital Olomouc, Olomouc, Czechia
  - Institute for the Care of Mother and Child, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No